CLINICAL TRIAL: NCT04488263
Title: Natural History Study of Children and Adults With Neuroendocrine Neoplasms (NENs)
Brief Title: Natural History Study of Children and Adults With Neuroendocrine Neoplasms (NEN)s
Status: Terminated | Type: Observational
Why Stopped: To avoid the duplication of effort and resources associated with the PI's branch change.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200139; 20-C-0139
Record Dates: First submitted 2020-07-24; First posted 2020-07-27 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Neuroendocrine Tumors; Carcinoma, Neuroendocrine
Keywords: Clinical Outcome; Advice in the Management of Cancer; Patterns of Disease Progression; Response or Lack of Response to Therapeutic Interventions; Natural History
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Subjects with confirmed/suspected NENs.

SUMMARY:
Background:

Neuroendocrine neoplasms (NENs) are rare tumors that originate in neuroendocrine cells. NENs can affect almost any part of the body. People with low-grade tumors can live many years. But high-grade tumors can be very aggressive. Researchers want to learn more about this type of cancer. This may help them design better treatments and supportive care studies.

Objective:

To gain a better understanding of neuroendocrine neoplasms.

Eligibility:

People starting at age 3 and older who have or are suspected of having NENs and are enrolled in protocol 19C0016, Natural History and Biospecimen Acquisition Study for Children and Adults with Rare Solid Tumors

Design:

Participants will be screened with questions about their medical history. This may be done over the telephone or in person.

Participants medical records, test results, and imaging results will be reviewed. They may have scans and blood tests. They may sign a separate consent form for some of the tests.

Participants will complete paper or electronic surveys. The surveys will ask about the effects of cancer on their wellbeing.

Participants may give samples of their tumors from previous surgeries or biopsies. These samples will be used to study their tumor genes.

Participants will get advice on how to manage their NENs. They will also get recommendations about potential treatment options.

Participants home doctors will be contacted every 6 to 12 months. They will give medical data such as imaging and test results.

Participants may have follow-up visits at NIH every 6 to 12 months.

Participants will contact researchers if there are any changes in their tumor.

Participants will be followed on this study for life.

DETAILED DESCRIPTION:
Background:

* Neuroendocrine neoplasm (NENs) are divided into neuroendocrine tumors (NETs) and neuroendocrine carcinomas (NECs). These are rare malignancies occurring for example in the gastrointestinal tract, islets of the pancreas, lung, adrenal medulla, thyroid C-cells, etc. and are heterogeneous group of neoplasms with unique tumor biology, natural history, and clinical management issues.
* Their incidence has increased over the last decade, with an incidence of 6 per 100,000 persons a year and they represent 0.46% of all malignancies.
* Most NETs are sporadic, but they can be part of familial cancer syndromes such as multiple endocrine neoplasia type 1 (MEN1), neurofibromatosis type 1 (NF1) or Von Hippel- Lindau (VHL) syndrome. Whereas poorly differentiated neuroendocrine carcinomas (NECs) are all high-grade carcinomas that resemble small cell carcinoma or large cell carcinoma of the lung.
* Treatment for localized NETs is surgical resection, however, a variety of therapeutic options are available for patients with advanced NETs. When to apply a given option, what combination therapeutic approach should be used, how long treatment should be continued should be used is unclear and controversial.

Objective:

-Characterize the natural history of neuroendocrine neoplasms (NENs). Data will include clinical presentation, patterns of disease progression, response or lack of response to therapeutic interventions, disease recurrence and overall survival.

Eligibility:

* Subjects with confirmed or suspicion of NENs.
* Age greater than or equal to 3 years old

Design:

* This protocol is a subprotocol of protocol 19C0016 Natural History and Biospecimen Accrual Study for Children and Adults with Rare Solid Tumors . After enrollment on the master protocol and undergoing evaluations detailed in the master protocol, patients will be enrolled on this subprotocol specific for NENs.
* Medical histories will be documented, and patients followed throughout the course of their illnesses, with particular attention to patterns of disease recurrence and progression, response to therapies, duration of responses and hormone production in patients with hormone production as a manifestation of their disease. Tumor growth rates will also be calculated throughout the course of the disease.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Enrollment into NCI protocol 19C0016 'Natural History and Biospecimen Acquisition Study for Children and Adults with Rare Solid Tumors'.
* Age greater than or equal to 3 years old
* Ability of subject or parent/guardian to understand and the willingness to sign a written consent document.
* Subjects with:

  --histologically or cytologically documented NENs, OR
* biochemical evidence of neuroendocrine tumor (serum/urinary) based on elevated levels of chromogranin A, pancreatic polypeptide, neuron-specific enolase, vasoactive intestinal polypeptide, serotonin (urinary 5-HIAA), gastrin, somatostatin, catecholamines, metanephrines, calcitonin, fasting insulin, C-peptide (proinsulin), glucagon, anterior pituitary hormones, OR
* Suspicion of NEN (from any site/origin) on axial imaging (CT/MRI/FDG, PET/68Ga-DOTATATE scan, FDOPA PET scan).

EXCLUSION CRITERIA:

None

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
natural history of neuroendocrine neoplasms | ongoing
  clinical presentation, patterns of disease progression, response or lack of response to therapeutic interventions, disease recurrence and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jaydira Del Rivero, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0139.html